CLINICAL TRIAL: NCT00379860
Title: A Multiple Ascending Dose Study of the Safety, Pharmacokinetics, and Pharmacodynamics of LXR-623 Administered Orally to Healthy Subjects
Brief Title: Study Evaluation LXR-623 in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3201A1-101
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2007-03-09 (Estimated); Status verified 2007-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — 2-(2-chloro-4-fluorobenzyl)-3-(4-fluorophenyl)-7-(trifluoromethyl)-2H-indazole

INTERVENTIONS:
Drug: LXR-623

SUMMARY:
To evaluate the safety and tolerability of multiple doses of LXR in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy adults.
* Liver function tests, triglycerideres, and creatinine must be below upper limit of normal at screening.

Exclusion Criteria:

* A history or active presence of clinically important medical disease.
* Any metal implants or devices.
* Claustrophobia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-10; Study Completion 2007-01

PRIMARY OUTCOMES:
Safety is the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer